CLINICAL TRIAL: NCT06423599
Title: Effect of Weight Loss on Physical and Cardiac Performance in People With Obesity and Heart Failure
Acronym: FIT-HF
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jens D Hove, MD,PHD (Other)
Responsible Party: Sponsor-Investigator, Jens D Hove, MD,PHD, Chief Physician, Research associate Professor, MD, PhD, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1298-6418; 2023-503753-35-01 (EU CTIS Number)
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Obesity; Weight Loss; Chronic Heart Failure
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: This is a investigator-initiated, parallel-group, 2-arm assessor-blinded, open-label, randomised, clinical trial
Who Masked: Outcomes Assessor
Masking Description: Anonymized data will be analyzed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide intervention group (Experimental): Dose-escalation of semaglutide will take place during the first 16 weeks after randomisation (week 0). Patients will start at the 0.25 mg once-weekly dose and follow dose-escalation schedule (0.25, 0.5, 1.0, 1.7 and 2.4 mg). For all subjects we aim at reaching the recommended target dose of 2.4 mg semaglutide once weekly for the rest of the period of total 52 weeks.
  Interventions: Drug: Semaglutide Injectable Product
- Calorie-restricted diet intervention group (Active Comparator): In short, the weight loss program in the calorie-restricted diet group consists of 3 phases after randomisation (week 0). An initial weight loss phase of 8 weeks with 800 calories/day, a food re-introduction phase for 8 weeks and a weight loss maintenance phase for the rest of the period of total 52 weeks.
  Interventions: Dietary Supplement: Calorie-restricted diet

INTERVENTIONS:
Drug: Semaglutide Injectable Product — Weight loss using Semaglutide
  Arms: Semaglutide intervention group
Dietary Supplement: Calorie-restricted diet — Weight loss by calorie-restricted diet program followed by a weight loss maintenance follow-up program
  Arms: Calorie-restricted diet intervention group

SUMMARY:
The benefit of weight loss in patients with obesity and heart failure with reduced ejection fraction (HFrEF) is controversial. Semaglutide has shown cardiovascular (CV) risk-reduction and impact on CV risk factors including overweight, dysglycaemia and hypertension in subjects with type 2 diabetes (T2D). The STEP-HFpEF (Semaglutide Treatment Effect in People With Obesity and HFpEF) recently demonstrated, at 1-year, to not only reduce weight considerably, but also significantly improve health-related quality of life, functional status scores and 6-min walk distance in patients with heart failure with preserved ejection fraction (HFpEF). Also, the recently concluded SELECT trial was the first CV outcome trial with semaglutide in patients with overweight or obesity and established CV disease, including heart failure (but no T2D). Semaglutide demonstrated a 20% reduction in MACE, defined as the composite of cardiovascular death, non-fatal myocardial infarction, and non-fatal stroke.

These landmark findings have important implications for clinicians -as they mean that weight loss and/or semaglutide as anti-obesity pharmacotherapy could be a treatment strategy for secondary prevention of CV disease in patients with overweight or obesity.

It is, however, unknown whether weight loss with either calorie-restricted diet or semaglutide has beneficial effects in obese subjects with heart failure and reduced ejection fraction. Also it is unclear whether semaglutide has cardiovascular benefits irrespective of starting weight and amount of weight loss.

Purpose: The study aims to investigate whether weight loss treatment with semaglutide is superior to weight loss with calorie-restricted diet in improving peak oxygen uptake in patients with obesity and heart failure with reduced ejection fraction.

DETAILED DESCRIPTION:
Background: The prevalence of overweight and obesity has reached pandemic proportions. Obesity is known to increase the risk for Type 2 diabetes and hypertension, as well as the risk for overt cardiovascular (CV) disease, including myocardial infarction, heart failure, and stroke. The rising prevalence of obesity may counteract the recent advances in primary and secondary prevention of CV disease. Overweight and obesity are common in patients with CV disease; however, cardiologists face several challenges in managing body weight in this population. Many may not consider obesity as a therapeutic target probably because there were no previous highly effective and safe pharmacologic interventions to consider. In addition, they may not have the expertise or resources to implement lifestyle interventions and may have limited familiarity with obesity pharmacotherapy. Moreover, the long-term CV effects of obesity pharmacotherapy remain uncertain due to limited CV outcome data with weight loss as the primary intervention. Although current CV guidelines recognize the importance of weight loss, they primarily focus on lifestyle modifications, with fewer details on strategies to utilize obesity pharmacotherapy and surgery. However, the recent 2022 American Diabetes Association/European Association for the Study of Diabetes consensus on the management of Type 2 diabetes has moved up weight management to the front of the treatment algorithm, by prioritizing the use of pharmacologic interventions such as glucagon-like peptide-1 receptor agonists and dual glucose-dependent insulinotropic polypeptide/glucagon-like peptide-1 receptor agonists, which have potent weight-lowering effects, in addition to glucose-lowering effects.

Hypothesis: The investigators hypothesise that weight loss treatment with semaglutide is superior to weight loss with state-of-the-art calorie-restricted diet in improving the peak oxygen uptake (ml/min/kg) after 52 weeks as a marker of physical performance (and with prognostic implications) in patients with obesity and heart failure with reduced ejection fraction.

Design: This is a investigator-initiated, parallel-group, 2-arm assessor-blinded, open-label, randomised, controlled trial (RCT) comparing the effect of weight loss using low-calorie replacement diet to weight loss using semaglutide in obese patients with heart failure with reduced ejection fraction. Subjects will be randomised in a 1:1 ratio to receive either low-calorie replacement diet or semaglutide.The subjects wil be followed for 52 weeks during the intervention period. The patients will be examined at 16 weeks (where the weight loss is anticipated to be approximately equal in the two groups) and after 52 weeks.

Primary, secondary and exploratory objectives are listed below. The exploratory objectives are mostly embedded mechanistic studies of an exploratory nature and therefore hypothesis-generating in the RCT.

Intervention: Subjects will be treated with semaglutide once weekly or a weight loss intervention consisting of a calorie-restricted diet and dietary advice on top of standard of care, which covers management of heart failure medication, CV risk factors and healthy lifestyle counselling.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years at the time of signing informed consent
* Body mass index (BMI) ≥ 30 kg/m2
* Heart failure with New York Heart Association (NYHA)-class 1-3 and reduced ejection fraction (EF≤40%) established by either:

  1. echocardiography AND/OR
  2. cardiac magnetic resonance
* On stable optimal medical heart failure therapy for at least 4 weeks

Exclusion Criteria:

1. Cardiovascular-related:

   * Any of the following: myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within the past 6 months prior to the day of screening
   * Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
   * Transient heart failure related to reversible mechanisms like tachycardia, sepsis, etc.
2. Glycaemia-related:

   * Type 1 diabetes
   * Treatment with any Glucagon-Like Peptide-1 (GLP-1) agonists within 90 days prior to the day of screening
   * Type 2 diabetes requiring other pharmacotherapy than metformin and Sodium-glucose Cotransporter-2 (SGLT2) Inhibitors
3. General safety:

   * Pregnancy or planned pregnancy
   * History or presence of chronic pancreatitis
   * Presence of acute pancreatitis within the past 180 days prior to the day of screening
   * Kidney disease with eGFR < 35ml/min
   * Presence or history of malignant neoplasms within the past 5 years prior to the day of screening (Basal and squamous cell skin cancer and any carcinoma in-situ are allowed)
   * Known or suspected hypersensitivity to trial product(s) or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen uptake | The patients will be examined after 0, 16 and 52 weeks
  To examine the effect of weight loss on mean change in peak oxygen uptake at 52 weeks between semaglutide and calorie-restricted group compared to baseline (Measured in ml O2/(kg x min))

SECONDARY OUTCOMES:
The Clinical Summary Score of the Kansas City Cardiomyopathy Questionnaire (KCCQ-CSS) | The patients will be examined after 0, 16 and 52 weeks.
  To compare the effect of weight loss on the mean change
6-min walk distance (6MWD) | The patients will be examined after 0, 16 and 52 weeks
  To compare the effect of weight loss on the mean change
End-systolic volume of the left ventricle assessed by Cardiac MRI | The patients will be examined after 0, 16 and 52 weeks
  To compare the effect of weight loss on the mean change
N-terminal pro-B-type natriuretic peptide (NT-proBNP) and C-reactive protein (CRP) change | The patients will be examined after 0, 16 and 52 weeks
  To compare the effect of weight loss on the mean change

OTHER OUTCOMES:
Composite endpoint consisting of all-cause death, non-fatal myocardial infarction, non-fatal stroke, heart failure hospitalisation or urgent heart failure visit | Follow-up at 52 weeks
First occurrence of a composite heart failure endpoint consisting of: heart failure hospitalisation, urgent heart failure visit, ischemic events or CV death | Follow-up at 52 weeks
All-cause death | Follow-up at 52 weeks
Total number of hospitalised days | Follow-up at 52 weeks
Total number of hospitalisations | Follow-up at 52 weeks
Total number of Serious Adverse Events (SAEs) | Follow-up at 52 weeks
Change in heart failure medication | Follow-up at 52 weeks
EuroQol five dimensions five level (EQ-5D-5L) questionnaire | The patients will answer a questionnaire after 0, 16 and 52 weeks
  To examine the effect of a weight loss with either calorie-restricted diet or semaglutide on quality of life in patients with obesity and heart failure with reduced EF
Effects of weight loss with either treatment on cardiac metabolism, fibrosis, inflammation, and diastolic function by Cardiac MRI and Cardiac Rubidium-PET | The patients will be examined after 0, 16 and 52 weeks
Potentially favorable changes in other organ systems caused by weight loss in this patient group | The patients will be examined after 0, 16 and 52 weeks
  Analysis of: Blood samples, pulmonary function test and body composition scan (DEXA)
Feasibility and safety of two modern weight loss programs for aggressive weight lowering in patients with heart failure with reduced ejection fraction. | Follow-up at 52 weeks
Changes in systolic and diastolic function and cardiac morphology assessed by echocardiography | The patients will be examined after 0, 16 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jens D Hove, Principal Investigator — Amager-Hvidovre Universitetshospital
Locations (1):
- Amager and Hvidovre Hospital University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No